CLINICAL TRIAL: NCT01997190
Title: A Phase I Study of Intrapleural AdV-tk Therapy in Patients With Malignant Pleural Effusion
Brief Title: Intrapleural AdV-tk Therapy in Patients With Malignant Pleural Effusion
Acronym: MpeTK01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MpeTK01
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Malignant Pleural Effusion; Lung Cancer; Mesothelioma; Breast Cancer; Ovarian Cancer
Keywords: Immunotherapy; Gene therapy; Tumor vaccine
MeSH Terms: conditions — Pleural Effusion, Malignant; Lung Neoplasms; Mesothelioma; Breast Neoplasms; Ovarian Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Arm (Experimental): AdV-tk + valacyclovir
  Interventions: Biological: AdV-tk + valacyclovir

INTERVENTIONS:
Biological: AdV-tk + valacyclovir — AdV-tk will be administered intrapleural through pleural catheter followed by oral valacyclovir. Valacyclovir will be administered orally at a fixed dose for 14 days after each AdV-tk administration.

SUMMARY:
This is a phase I study of intrapleural AdV-tk therapy in patients with malignant pleural effusion (MPE). The primary objective is to test the safety of intrapleural AdV-tk therapy. Secondary objectives are to evaluate clinical efficacy and biologic activity

DETAILED DESCRIPTION:
The goal of this open-label, dose escalation clinical trial is to investigate if the administration of AdV-tk to patients with MPE followed by valacyclovir and chemotherapy is safe, can be effectively delivered without disturbing standard therapy, and will have anti-tumor activity in patients with solid tumors.

The first and second dose levels have been completed, and the study is currently expanded to enroll more patients to dose level 2 with Celecoxib.

Patients will receive one injection of AdV-tk through a pleural catheter on day 0. The prodrug, valacyclovir, will be administered orally at a fixed dose for 14 days after each AdV-tk injection. Celecoxib will be administered starting 3 days before AdV-tk and continuing for 2 days after AdV-tk administration.

Chemotherapy may begin at any time after completion of valacyclovir. Choice of chemotherapy depends on the treating oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have MPE (defined as positive pleural fluid cytology). Eligible patients include NSCLC, small cell lung cancer, malignant mesothelioma (MM), breast cancer and ovarian cancer. Diagnosis must be made prior to AdV-tk injection. For patients with MM, histologic proof is needed, but positive pleural fluid cytology is not required.
* Patients must have an indication for placement of pleural catheter
* Patients must be 18 years of age or older
* Performance status must be ECOG 0-1
* Acute toxic effects from any prior radiotherapy, chemotherapy, or prior surgical procedures must have resolved to NCI CTCAE v 4.0 grade ≤ 1
* Baseline pulmonary function tests must be FEV1 ≥1 liter or 40% of predicted value (may be post-drainage and/or bronchodilator)
* Bilirubin ≤ 1.5 x upper limit of normal (ULN) and ALT, AST and alkaline phosphatase ≤ 2 x ULN
* Serum creatinine < 2 mg/dl and calculated creatinine clearance > 30 ml/min
* Hemoglobin ≥ 9 g/dL, ANC > 1000/mm3 and platelets > 100,000/mm3
* Serum albumin level ≥ 2.5 g/dL
* Patients must give study specific informed consent prior to enrollment

Exclusion Criteria:

* Patients may not be on systemic corticosteroids (>10 mg prednisone per day) or other systemic immunosuppressive drugs
* Patient is not known to be HIV+
* Patient is not pregnant or breast-feeding. Female patients of childbearing age must have negative serum or urine pregnancy test within 1 week of beginning therapy.
* Patient may not have clinically significant pericardial effusion
* Patient may not have other serious co-morbid illness or compromised organ function
* Patient may not have liver disease including known cirrhosis, active hepatitis or chronic active hepatitis B
* No prior allergic reaction or hypersensitivity to sulfonamides, celecoxib, aspirin or other NSAIDs
* No concurrent use of other NSAID or aspirin exceeding 100mg/day during celecoxib administration. No wash-out period required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 8 weeks

SECONDARY OUTCOMES:
Progression-free survival | 5 years
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aggarwal C, Haas AR, Metzger S, Aguilar LK, Aguilar-Cordova E, Manzanera AG, Gomez-Hernandez G, Katz SI, Alley EW, Evans TL, Bauml JM, Cohen RB, Langer CJ, Albelda SM, Sterman DH. Phase I Study of Intrapleural Gene-Mediated Cytotoxic Immunotherapy in Patients with Malignant Pleural Effusion. Mol Ther. 2018 May 2;26(5):1198-1205. doi: 10.1016/j.ymthe.2018.02.015. Epub 2018 Feb 21. PMID 29550074
- See also: Phase I Study of Intrapleural Gene-Mediated Cytotoxic Immunotherapy in Patients with Malignant Pleural Effusion — https://pubmed.ncbi.nlm.nih.gov/29550074/